CLINICAL TRIAL: NCT02031172
Title: Effects of Sustained Reading on the Ocular Surface
Status: Terminated | Type: Observational
Why Stopped: PI is moving to a different institution.
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Holly Hindman, Assistant Professor, University of Rochester
Other Study IDs: 00048640
Record Dates: First submitted 2013-12-02; First posted 2014-01-09 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Dry Eye Syndromes; Sjogren's Syndrome
Keywords: Dry Eye Disease; Sjogren's Syndrome; Tear Film; Ocular Surface; Aqueous Tear Deficiency
MeSH Terms: conditions — Dry Eye Syndromes; Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Subjects with Dry Eye Disease: Measures tear film stability, and visual function will be taken before and after a sustained silent reading task. The reading task will take place over 30 minutes, and a comprehension assessment will be given after reading. After completion of the reading task, measures of corneal sensation and structural imaging will be performed. The results from each of 3 cohorts will be compared to ascertain the differences between those populations with and without dry eye.
- Subjects with Sjogren's Syndrome: Measures tear film stability, and visual function will be taken before and after a sustained silent reading task. The reading task will take place over 30 minutes, and a comprehension assessment will be given after reading. After completion of the reading task, measures of corneal sensation and structural imaging will be performed. The results from each of 3 cohorts will be compared to ascertain the differences between those populations with and without dry eye.
- Healthy Controls: Measures tear film stability, and visual function will be taken before and after a sustained silent reading task. The reading task will take place over 30 minutes, and a comprehension assessment will be given after reading. After completion of the reading task, measures of corneal sensation and structural imaging will be performed. The results from each of 3 cohorts will be compared to ascertain the differences between those populations with and without dry eye.

SUMMARY:
This research is being done to to see if changes in visual reading function correlate with changes in optical and retinal image quality. We hypothesize that changes and deterioration in tear film quality and dynamics may have a negative effect on reading function.

People with or without dry eye syndrome may enroll.

ELIGIBILITY:
General inclusion criteria for all subjects will include:

* Ages 50 to 89 years
* Capacity to give informed consent.
* Self-reported literacy (i.e. a "Yes" answer to the question "Have you learned how to read?")

Additional inclusion criteria for the dry eye group will include both of the below:

* A previous diagnosis of dry eye syndrome by an eyecare specialist
* Ocular Surface Disease Index total scoring of 13 or above

Additional inclusion criteria for the Sjögren's syndrome group will include:

- A previous diagnosis of Sjögren's syndrome by an immunology specialist, per ACR criteria 22

Additional inclusion criteria for normal control subjects will include:

* No previous history of dry eye diagnosis
* Ocular Surface Disease Index total scoring of 12 or under
* Total corneal and conjunctival staining score of 0

Exclusion criteria will include:

* A binocular vision below 20/25 (with habitual correction)
* Any ocular surgery within the last 3 months.
* Mental issues, illiteracy, or language problems which might possibly interfere with reading ability
* History of taking or current use of topical prescription anti-inflammatory eyedrops (including, cyclosporine and steroids as well as any glaucoma eyedrops). Subjects who are willing to discontinue their treatment for at least a period of 30 days can be placed on a "wash out period" as per the discretion of the investigator and subject safety, and be eligible at the end of this period, given all other criteria have been met. Otherwise, subjects on these medications will be excluded.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We plan to recruit 50 subjects from 3 populations (dry eye, Sjogren's, and healthy controls). Subjects will be recruited regardless of gender, race, or ethnicity; and enrollment will based on specific criteria as described below.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2014-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
To see if changes in visual reading function correlate with changes in optical and retinal image quality, secondary to changes in tear film dynamics | 30 minutes
To determine whether corneal sensation and corneal nerve morphology correlate with sustained reading function | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Holly B Hindman, MD, Principal Investigator — University of Rochester, Flaum Eye Institute
Locations (1):
- University of Rochester, Rochester, New York, United States